CLINICAL TRIAL: NCT06108843
Title: Effects of the Myofascial Arm Pull With and Without Active Release Technique on Pain, Range of Motion and Disability in Adhesive Capsulitis
Brief Title: Effects of the Myofascial Arm Pull With and Without Active Release Technique in Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0162
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Active Release Technique; Myofacial Arm Pull Technique; Pain; Range of Motion
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Intervention Model Description: A type of intervention model describing a clinical trial in which two or more groups of participants receive different interventions.
Who Masked: Participant
Masking Description: A participant in a single-blind study does not know which study group they are in, but the study doctor does.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial arm pull technique and Active Release Technique (Experimental): Participant will receive both Myofascial arm pull and active release technique along with Ultrasound therapy.
  Interventions: Other: Myofascial Arm Pull and Active Release Technique
- Myofascial arm pull technique (Active Comparator): Participant will receive Myofascial arm pull along with ultrasound therapy.
  Interventions: Other: Myofacial Arm Pull

INTERVENTIONS:
Other: Myofascial Arm Pull and Active Release Technique — Six weekly sessions of the treatment will be given over the course of four weeks. Baseline treatment includes Ultrasound for 10 minutes.
  Arms: Myofascial arm pull technique and Active Release Technique
Other: Myofacial Arm Pull — Six weekly sessions of the treatment will be given over the course of four weeks. Baseline treatment includes Ultrasound for 10 minutes.
  Arms: Myofascial arm pull technique

SUMMARY:
The aim of the study is to determine the effects of the myofascial arm pull with and without active release technique on pain, ROM and disability in adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis (frozen shoulder), a painful disorder caused by capsular inflammation that results in fibrosis and rigidity of the glenohumeral joint capsule, is characterized by a progressive loss of both active and passive glenohumeral movements. Frozen shoulder can be primary (also known as idiopathic) if there is no underlying cause of disease or it can be secondary. The term "secondary frozen shoulder" is associated with injury, trauma, cardiovascular diseases, hemiparesis, or diabetes.Active release technique and myofascial arm pull technique are both effective treatment options for patients with adhesive capsulitis. These techniques help to improve range of motion and reduce pain by releasing tension and adhesions in the affected area. Active release technique focuses on releasing tension and adhesions in the soft tissues surrounding the affected joint, while the Myofascial arm pull technique aims to improve range of motion by stretching the muscle and fascia in the affected area. By incorporating these techniques into a comprehensive treatment plan, patients of adhesive capsulitis can see significant improvement in their pain, range of motion and disability.

Because the method of treatment is inexpensive, findings of this study could be beneficial in revision of the clinical protocols to manage the patients of adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female; mean age (35-60).
* Case diagnosed with adhesive capsulitis, both primary and secondary origin.
* Freezing stage of adhesive capsulitis.
* Those with at least a 50% reduction in the range of motion (ROM).

Exclusion Criteria:

* History of shoulder surgery or manipulation under anesthesia, local corticosteroid injection administration to the affected shoulder within the last 3 months.
* Neurological deficit affecting the shoulder functioning during daily activities.
* Pathology of the shoulder joint other than adhesive capsulitis.
* Pain or disorder of the cervical spine, elbow, wrist or hand.
* Patients diagnosed with cancer

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and disability index (SPADI) | 4 week
  Changes from Baseline. The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability
Goniometer | 4 week
  Changes from Baseline. Physical therapists use goniometry to objectively measure passive and active range of motion (ROM).
Numeric Pain Rating Scale (NPRS) | 4 week
  Changes from Baseline. The NPRS is a self-reported, or clinician administered, measurement tool The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10.
  0=No pain
  1 to 4=Mild pain. 5 or 6=Moderate pain 7 to 10=Severe pain

CONTACTS AND LOCATIONS:
Overall Officials: FAIZA AMJAD, M.PHILL, Principal Investigator — Riphah International University
Locations (1):
- Arif Memorial Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogru H, Basaran S, Sarpel T. Effectiveness of therapeutic ultrasound in adhesive capsulitis. Joint Bone Spine. 2008 Jul;75(4):445-50. doi: 10.1016/j.jbspin.2007.07.016. Epub 2008 May 2. PMID 18455944
- [Background] Sumariva-Mateos J, Leon-Valenzuela A, Vinolo-Gil MJ, Bautista Troncoso J, Del Pino Algarrada R, Carmona-Barrientos I. Efficacy of myofascial therapy and kinesitherapy in improving function in shoulder pathology with prolonged immobilization: A randomized, single-blind, controlled trial. Complement Ther Clin Pract. 2022 Aug;48:101580. doi: 10.1016/j.ctcp.2022.101580. Epub 2022 Apr 4. PMID 35397306
- [Background] Breckenridge JD, McAuley JH. Shoulder Pain and Disability Index (SPADI). J Physiother. 2011;57(3):197. doi: 10.1016/S1836-9553(11)70045-5. PMID 21843839
- [Background] Angst F, Goldhahn J, Pap G, Mannion AF, Roach KE, Siebertz D, Drerup S, Schwyzer HK, Simmen BR. Cross-cultural adaptation, reliability and validity of the German Shoulder Pain and Disability Index (SPADI). Rheumatology (Oxford). 2007 Jan;46(1):87-92. doi: 10.1093/rheumatology/kel040. Epub 2006 May 23. PMID 16720638
- [Background] Mullaney MJ, McHugh MP, Johnson CP, Tyler TF. Reliability of shoulder range of motion comparing a goniometer to a digital level. Physiother Theory Pract. 2010 Jul;26(5):327-33. doi: 10.3109/09593980903094230. PMID 20557263
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114